CLINICAL TRIAL: NCT04233359
Title: Local Anesthetic Thoracoscopy Versus Ultrasound Guided Pleural Biopsies and Repeat Thoracocentesis in Pleural Effusion After Inconclusive Initial Thoracentesis: a Randomized Study
Brief Title: A Randomised Study Evaluating Diagnostics of Pleural Effusion Among Patients Suspect of Cancer.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To few patients recruited to allow for study completion within ph.d. project.
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-790
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pleural Effusion, Malignant; Pleural Effusion; Pleura; Exudate
Keywords: Pleural effusion; Malignant Pleural effusion; Pleura diagnostics; US-guided pleural biopsy; Local anesthetic thoracoscopy
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided pleural biopsy and thoracentesis (Active Comparator): Pleural biopsy:
  Using ultrasound the optimal point of entry for thoracentesis is located, and local anesthesia is obtained. The area is wiped with disinfectant and a skin incision is made with a pointed scalpel. Six US-guided biopsies of 1x2 millimetres are taken from the parietal pleura using closed needle biopsies (Quick-core Biopsy Needle 18G, COOK Medical, Bloomington, Indiana, USA or Bard Max Core Biopsy Needle 18G, Tempe, Arizona, USA). Afterward, a thoracentesis is performed in the same incision as used by the pleural biopsy. A pigtail catheter is inserted and fastened and connected to a sealed bag and fluid is aspirated and sent to relevant analysis.
  Interventions: Procedure: US-guided pleural biopsy
- LAT and thoracentesis (Experimental): Local anesthetic thoracoscopy: Pre-procedure a pleural pigtail catheter is inserted and pleural fluid is removed. The catheters one-way valve is opened and the patient takes several breaths thereby creating a pneumothorax prior to procedure start. The patient is sedated with midazolam and morphine. Midaxillary access through intercostal space 4-7 is achieved in local anesthesia and via a skin incision a trocar is placed for access to the thoracic space. A semi-rigid thoracoscope (model LTF 160; Olympus, Tokyo, Japan) is inserted via the trocar and the pleural cavity is inspected after removal of residual effusion whereof at least 40ml is sent to cytology. Pleural parietal biopsies are taken under direct visual guidance. The recommended number of biopsies is 10-15. If no abnormalities were seen, random biopsies are taken. After relevant biopsies are taken the instruments are removed the pigtail catheter stays inserted to allow for removal of air and expansion of the lung.
  Interventions: Procedure: Local anesthetic thoracoscopy

INTERVENTIONS:
Procedure: Local anesthetic thoracoscopy — Procedure to obtain histological biopsies of the parietal pleura on awake, fastening patients.
  Other Names: medical thoracoscopy
  Arms: LAT and thoracentesis
Procedure: US-guided pleural biopsy — In local anesthesia, a closed needle biopsy is performed Ultrasound guided of the parietal pleura at the place of deepest fluid recess in the intrathoracic space. A pigtail catheter French 7-16 is placed afterwards for fluid drainage.
  Arms: US-guided pleural biopsy and thoracentesis

SUMMARY:
Pleural fluid can be caused by cancer. Patients with repeated presentation of pleural fluid where initial diagnostic tests have been inconclusive are the focus of this trial. In this clinical trial patients are randomized into two groups and the efficacy of local anesthetic thoracoscopy (LAT) is compared to an ultrasound guided biopsy of the outer lining of the lung. The aim is not only the diagnostic yield in diagnosing cancer, but also the procedures ability to diagnose specific cancer mutations and immune system markings.

Methods and objectives:

Patients with reoccuring one-sided pleural fluid, with a marked clinical risk of cancer based on findings in medical work-up, radiological scans, biochemistry and medical history and who are undiagnosed upon initial pleural fluid analysis are the target patients of the trial. Patients are randomized into two groups to have undertaken either pleural biopsy at the optimal site for a repeat thoracentesis or LAT. Thus diagnostic yield for both fluid analysis and biopsy analysis will be compared to tissue samples taken with LAT.

We hypothesize that LAT is superior both to pleural biopsy and repeat thoracentesis in providing diagnostic clarification and providing sufficient basis for treatment without further procedures resulting in less time consumption, cost and discomfort for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older patients with single previous thoracentesis of a unilateral pleural exudate according to Lights criteria without malignant cells.
* Lights Criteria:

Pleural fluid protein/serum protein ratio greater than 0.5 pleural fluid LDH/serum LDH ratio greater than 0.6 Pleural fluid LDH greater than two-thirds the upper limits of the Laboratorys normal Serum LDH

* Contrast enhanced CT of the Chest and abdomen performed
* Clinical suspicion of cancer such as, but not limited to, weight loss, malaise, anemia
* Pet-CT results or former cancer diagnosis Informed consent

Exclusion Criteria:

* bilateral pleural effusions
* known cause of pleural effusion
* likely non-malignant course of a unilateral pleura effusion such as (but not restricted to) pneumonia, trauma, pleuritis, heart failure
* any contraindication to the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-guiding pleural workup to provide and plan treatment for the cause of the pleura exudate, local anesthetic thoracoscopy vs 2. thoracentesis | 26 weeks
  Difference in incidence of treatment-guiding diagnostic workup in local anesthetic thoracoscopy versus 2nd thoracentesis
Incidence of treatment-guiding pleural workup to provide and plan treatment for the cause of the pleura exudate. Local anesthetic thoracoscopy vs US-guided pleural biopsy. | 26 weeks
  Difference in incidence of treatment-guiding diagnostic workup in local anesthetic thoracoscopy versus US-guided pleural biopsy prior to 2nd thoracentesis

SECONDARY OUTCOMES:
Incidence of achieving pleural immunohistochemistry, mutations, oncodrivers, culture and biochemistry. | 26 weeks
Incidence of completed procedures | 1 week
Time from randomization to conclusive, treatment-guiding diagnoses | 26 weeks
Time from start of consultation with medical staff until end of consultation with medical staff on the day of the procedure | Day of procedure/intervention
Time from procedure start to patient leaving the procedure room and leaving the recovery room | Day of procedure/intervention
Adverse event; complication to procedure: mortality | 30 days.
  Evaluated on day of procedure, 7 days and 30 days. The 2 last are performed via telephone call to the patient and informations gathering in the electronic patient file system
Adverse event; complication to procedure: pneumothorax | 30 days.
  Evaluated on day of procedure, 7 days and 30 days. The 2 last are performed via telephone call to the patient and informations gathering in the electronic patient file system
Adverse event; complication to procedure: haemoptysis | 30 days.
  Evaluated on day of procedure, 7 days and 30 days. The 2 last are performed via telephone call to the patient and informations gathering in the electronic patient file system
Adverse event; complication to procedure: infection | 30 days.
  Evaluated on day of procedure, 7 days and 30 days. The 2 last are performed via telephone call to the patient and informations gathering in the electronic patient file system
Adverse event; complication to procedure: hospital admission | 30 days.
  Evaluated on day of procedure, 7 days and 30 days. The 2 last are performed via telephone call to the patient and informations gathering in the electronic patient file system
Total volume of pleural fluid removed | Day of procedure
  In mililiter (ml)
Patient reported discomfort reported via ESAS | Day of procedure pre- and post-procedure and 1 week followup
  ESAS - Edmonton Symptom Assesment System, Danish Version 2008
Patient reported discomfort reported via EQ-5D-5L | Day of procedure pre- and post-proceudre and 1 week followup
  Denmark (Danish) © 2009 EuroQol Group EQ-5D™
Willingness to repeat procedure | After procedure performed - within 30 minutes and 1 week after proceudre
  5 Point Likert Scale, 1 not likely to repeat, 5 most likely to repeat
Cough | Pre-procedure, 1 week post procedure.
  Visual analogue scale 1-10. 1 Being no cough, 10 being extreme cough

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Bødtger, MD ph.d., Study Chair — Næstved
Locations (2):
- Denmark (2):
  - Næstved Hospital, Næstved
  - University Hospital Zealand, Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saks AM, Posner R. Tuberculosis in HIV positive patients in South Africa: a comparative radiological study with HIV negative patients. Clin Radiol. 1992 Dec;46(6):387-90. doi: 10.1016/s0009-9260(05)80684-1. PMID 1493651
- [Background] Arnold DT, De Fonseka D, Perry S, Morley A, Harvey JE, Medford A, Brett M, Maskell NA. Investigating unilateral pleural effusions: the role of cytology. Eur Respir J. 2018 Nov 8;52(5):1801254. doi: 10.1183/13993003.01254-2018. Print 2018 Nov. PMID 30262573
- [Background] Porcel JM, Esquerda A, Vives M, Bielsa S. Etiology of pleural effusions: analysis of more than 3,000 consecutive thoracenteses. Arch Bronconeumol. 2014 May;50(5):161-5. doi: 10.1016/j.arbres.2013.11.007. Epub 2013 Dec 20. English, Spanish. PMID 24360987
- [Background] Marel M, Zrustova M, Stasny B, Light RW. The incidence of pleural effusion in a well-defined region. Epidemiologic study in central Bohemia. Chest. 1993 Nov;104(5):1486-9. doi: 10.1378/chest.104.5.1486. PMID 8222812
- [Background] Bintcliffe OJ, Lee GY, Rahman NM, Maskell NA. The management of benign non-infective pleural effusions. Eur Respir Rev. 2016 Sep;25(141):303-16. doi: 10.1183/16000617.0026-2016. PMID 27581830
- [Background] Hooper C, Lee YC, Maskell N; BTS Pleural Guideline Group. Investigation of a unilateral pleural effusion in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii4-17. doi: 10.1136/thx.2010.136978. No abstract available. PMID 20696692
- [Background] Porcel JM, Gasol A, Bielsa S, Civit C, Light RW, Salud A. Clinical features and survival of lung cancer patients with pleural effusions. Respirology. 2015 May;20(4):654-9. doi: 10.1111/resp.12496. Epub 2015 Feb 23. PMID 25706291
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691
- [Background] Orki A, Akin O, Tasci AE, Ciftci H, Urek S, Falay O, Kutlu CA. The role of positron emission tomography/computed tomography in the diagnosis of pleural diseases. Thorac Cardiovasc Surg. 2009 Jun;57(4):217-21. doi: 10.1055/s-2008-1039314. Epub 2009 May 20. PMID 19670115
- [Background] Naito T, Satoh H, Ishikawa H, Yamashita YT, Kamma H, Takahashi H, Ohtsuka M, Hasegawa S. Pleural effusion as a significant prognostic factor in non-small cell lung cancer. Anticancer Res. 1997 Nov-Dec;17(6D):4743-6. PMID 9494600
- [Background] Nance KV, Shermer RW, Askin FB. Diagnostic efficacy of pleural biopsy as compared with that of pleural fluid examination. Mod Pathol. 1991 May;4(3):320-4. PMID 2068057
- [Background] Loddenkemper R, Boutin C. Thoracoscopy: present diagnostic and therapeutic indications. Eur Respir J. 1993 Nov;6(10):1544-55. PMID 8112449
- [Background] Garcia LW, Ducatman BS, Wang HH. The value of multiple fluid specimens in the cytological diagnosis of malignancy. Mod Pathol. 1994 Aug;7(6):665-8. PMID 7991525
- [Background] Koegelenberg CF, Irusen EM, von Groote-Bidlingmaier F, Bruwer JW, Batubara EM, Diacon AH. The utility of ultrasound-guided thoracentesis and pleural biopsy in undiagnosed pleural exudates. Thorax. 2015 Oct;70(10):995-7. doi: 10.1136/thoraxjnl-2014-206567. Epub 2015 May 21. PMID 25997433
- [Background] Light RW, Macgregor MI, Luchsinger PC, Ball WC Jr. Pleural effusions: the diagnostic separation of transudates and exudates. Ann Intern Med. 1972 Oct;77(4):507-13. doi: 10.7326/0003-4819-77-4-507. No abstract available. PMID 4642731
- [Background] Amiri Z, Momtahan M, Mokhtari M. Comparison of Conventional Cytology, Liquid-Based Cytology, and Cell Block in the Evaluation of Peritoneal Fluid in Gynecology Malignancies. Acta Cytol. 2019;63(1):63-72. doi: 10.1159/000495571. Epub 2019 Jan 9. PMID 30625466
- [Background] Pak MG, Roh MS. Cell-blocks are suitable material for programmed cell death ligand-1 immunohistochemistry: Comparison of cell-blocks and matched surgical resection specimens in lung cancer. Cytopathology. 2019 Nov;30(6):578-585. doi: 10.1111/cyt.12743. Epub 2019 Jul 19. PMID 31209979
- [Background] Metintas M, Yildirim H, Kaya T, Ak G, Dundar E, Ozkan R, Metintas S. CT Scan-Guided Abrams' Needle Pleural Biopsy versus Ultrasound-Assisted Cutting Needle Pleural Biopsy for Diagnosis in Patients with Pleural Effusion: A Randomized, Controlled Trial. Respiration. 2016;91(2):156-63. doi: 10.1159/000443483. Epub 2016 Jan 19. PMID 26779911
- [Background] Hallifax RJ, Corcoran JP, Ahmed A, Nagendran M, Rostom H, Hassan N, Maruthappu M, Psallidas I, Manuel A, Gleeson FV, Rahman NM. Physician-based ultrasound-guided biopsy for diagnosing pleural disease. Chest. 2014 Oct;146(4):1001-1006. doi: 10.1378/chest.14-0299. PMID 24832701
- [Background] Laursen CB, Naur TM, Bodtger U, Colella S, Naqibullah M, Minddal V, Konge L, Davidsen JR, Hansen NC, Graumann O, Clementsen PF. Ultrasound-guided Lung Biopsy in the Hands of Respiratory Physicians: Diagnostic Yield and Complications in 215 Consecutive Patients in 3 Centers. J Bronchology Interv Pulmonol. 2016 Jul;23(3):220-8. doi: 10.1097/LBR.0000000000000297. PMID 27454475
- [Background] Bibby AC, Dorn P, Psallidas I, Porcel JM, Janssen J, Froudarakis M, Subotic D, Astoul P, Licht P, Schmid R, Scherpereel A, Rahman NM, Maskell NA, Cardillo G. ERS/EACTS statement on the management of malignant pleural effusions. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):116-132. doi: 10.1093/ejcts/ezy258. PMID 30060030
- [Background] Feller-Kopman DJ, Reddy CB, DeCamp MM, Diekemper RL, Gould MK, Henry T, Iyer NP, Lee YCG, Lewis SZ, Maskell NA, Rahman NM, Sterman DH, Wahidi MM, Balekian AA. Management of Malignant Pleural Effusions. An Official ATS/STS/STR Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Oct 1;198(7):839-849. doi: 10.1164/rccm.201807-1415ST. PMID 30272503
- [Background] Willendrup F, Bodtger U, Colella S, Rasmussen D, Clementsen PF. Diagnostic accuracy and safety of semirigid thoracoscopy in exudative pleural effusions in Denmark. J Bronchology Interv Pulmonol. 2014 Jul;21(3):215-9. doi: 10.1097/LBR.0000000000000088. PMID 24992129
- [Background] Rozman A, Camlek L, Marc-Malovrh M, Triller N, Kern I. Rigid versus semi-rigid thoracoscopy for the diagnosis of pleural disease: a randomized pilot study. Respirology. 2013 May;18(4):704-10. doi: 10.1111/resp.12066. PMID 23418922
- [Background] Dhooria S, Singh N, Aggarwal AN, Gupta D, Agarwal R. A randomized trial comparing the diagnostic yield of rigid and semirigid thoracoscopy in undiagnosed pleural effusions. Respir Care. 2014 May;59(5):756-64. doi: 10.4187/respcare.02738. Epub 2013 Oct 8. PMID 24106326
- [Background] Rahman NM, Ali NJ, Brown G, Chapman SJ, Davies RJ, Downer NJ, Gleeson FV, Howes TQ, Treasure T, Singh S, Phillips GD; British Thoracic Society Pleural Disease Guideline Group. Local anaesthetic thoracoscopy: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii54-60. doi: 10.1136/thx.2010.137018. No abstract available. PMID 20696694
- [Background] Light RW. Diagnostic principles in pleural disease. Eur Respir J. 1997 Feb;10(2):476-81. doi: 10.1183/09031936.97.10020476. PMID 9042652
- [Background] Metintas M, Ak G, Dundar E, Yildirim H, Ozkan R, Kurt E, Erginel S, Alatas F, Metintas S. Medical thoracoscopy vs CT scan-guided Abrams pleural needle biopsy for diagnosis of patients with pleural effusions: a randomized, controlled trial. Chest. 2010 Jun;137(6):1362-8. doi: 10.1378/chest.09-0884. Epub 2010 Feb 12. PMID 20154079
- [Background] Swiderek J, Morcos S, Donthireddy V, Surapaneni R, Jackson-Thompson V, Schultz L, Kini S, Kvale P. Prospective study to determine the volume of pleural fluid required to diagnose malignancy. Chest. 2010 Jan;137(1):68-73. doi: 10.1378/chest.09-0641. Epub 2009 Sep 9. PMID 19741064
- [Background] Abouzgheib W, Bartter T, Dagher H, Pratter M, Klump W. A prospective study of the volume of pleural fluid required for accurate diagnosis of malignant pleural effusion. Chest. 2009 Apr;135(4):999-1001. doi: 10.1378/chest.08-2002. Epub 2008 Nov 18. PMID 19017891